CLINICAL TRIAL: NCT06104956
Title: Weaning Protocol for High-flow Nasal Oxygen Therapy in Intensive Care: A Multicentre Randomised Controlled Trial
Brief Title: Weaning Protocol for High-flow Nasal Oxygen Therapy in Intensive Care
Acronym: HiFloWEAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DR230001
Record Dates: First submitted 2023-10-12; First posted 2023-10-27 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Acute Hypoxemic Respiratory Failure; High-flow Nasal Oxygen Therapy
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group : Imposed weaning protocol (Experimental): The flow of the HFNO will remain high (50-60 L/min) guaranteeing the effectiveness of the HFNO on the wash-out of the anatomical space. At the same time, weaning will begin with a gradual reduction in FiO2 of 0.1 every 4 hours. To achieve this reduction, the patient will have to meet the safety targets of a stable respiratory rate at rest (no increase) and pulsed oxygen saturation (SpO2). The SpO2 target will be 92-95%. Once the FiO2 has stabilised at 0.4 for 4 hours, the nurse will initiate a 10 L/min reduction in the flow of HFNO every 4 hours. The oxygen therapy support may be changed for standard oxygen when the HFNO flow rate is 40L/min with an FIO2 of 0.4 for 4 consecutive hours.
  Interventions: Drug: HFNO weaning protocol
- Control group (Active Comparator): Weaning methods will be left to the free choice of the practitioner. Any change in the HFNO setting must be made on medical prescription. A minimum SpO2 objective is required (SpO2 ≥92%).
  Interventions: Drug: HFNO Standard of care

INTERVENTIONS:
Drug: HFNO weaning protocol — Algorithm based on SpO2 values and respiratory rate: a decrease of FiO2 and of the flow will be done
  Arms: Experimental group : Imposed weaning protocol
Drug: HFNO Standard of care — Weaning methods will be left to the free choice of the practitioner.
  Arms: Control group

SUMMARY:
High-flow nasal oxygen therapy (HFNO) is an oxygenation technique frequently used in intensive care.

The main objective of our study is to show that the use of a protocol for weaning patients off high-flow nasal oxygen therapy (HFNO) in the intensive care unit increases the probability that patients will be weaned from HFNO at Day 7 post-randomisation.

This is a open-label multicentre randomised controlled trial conducted in two parallel groups.

The primary endpoint is the success rate at Day 7, with success defined as "definitive" weaning from HFNO, i.e. patients weaned from HFNO for more than 48 hours without recourse to non-invasive ventilation (NIV) or intubation and still alive at Day 7.

The weaning protocol will be started as soon as the patient meets all the inclusion criteria, considered to be the prerequisites for initiating weaning from HFNO. Patients will be monitored until Day 28 maximum.

ELIGIBILITY:
Inclusion Criteria:

* Major patient admitted to the intensive care unit or continuous care unit for de novo hypoxaemic acute respiratory failure (with a PaO2/FiO2 ratio <300 mmHg)
* Treated with HDNO for at least 24 hours in an intensive care unit or continuous care unit
* Treated with HFNO with a flow rate ≥ 50L/min and inspired oxygen fraction (FiO2) ≥ 0.5, at inclusion
* With a ROX index (SpO2/FiO2/Respiratory Rate) stable or improving in the 6 hours prior to inclusion and greater than 4.88 (the patient must not be in a worsening phase).
* Had a blood gas test under HFNO within 24 hours of inclusion
* Participant covered by or entitled to social security
* Informed consent signed by the patient or its relatives if the patient is incapable; this consent must then be confirmed by the patient as soon as possible

Exclusion Criteria:

* Presence of a patient included in the study and not weaned off HFNO in the sector managed by the nurse of the patient assessed for eligibility
* Concomitant non-invasive ventilation treatment
* Use of HFNO within 7 days of extubation
* Chronic obstructive pulmonary disease (Gold grade 3 or 4)
* Cardiogenic acute pulmonary oedema as the main cause of acute respiratory failure
* Diffuse interstitial lung disease as a medical history
* Patient with long-term non-invasive ventilation with external positive pressure
* Patient on long-term oxygen therapy at home
* Pregnant women, women in labour and breastfeeding mothers
* Persons deprived of their liberty by a judicial or administrative decision, persons hospitalised without consent and persons admitted to a health or social establishment for purposes other than research.
* Minor
* Adult subject to a legal protection measure (guardianship, curators, person under court protection)
* Patient with a medical decision not to intubate
* Patients already included in the study, neither for the same stay if they were to present the inclusion criteria again, nor for subsequent stays

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2024-02-17 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The success rate at Day 7 | At day 7
  Success being defined as "definitive" weaning from HFNO, i.e. a patient weaned for more than 48 hours from HFNO without recourse to non-invasive ventilation or intubation and still alive at Day 7.

SECONDARY OUTCOMES:
High-flow nasal oxygen therapy (HFNO) weaning rate at day 28 | At day 28
Time to definitive weaning from HFNO | From randomisation to day 28
Cumulative incidence of intubation | From randomisation to day 28
Cumulative incidence of use of curative non-invasive ventilation | From randomisation to day 28
Mortality rate at day 28 | At Day 28
Number of days on HFNO for patients definitively weaned from HFNO | From randomisation to discharge from intensive care or at Day 28
Changes in the ROX index during the weaning phase | From randomisation to day 28
  ROX index : [(SpO2/FiO2)/respiratory rate]
Changes in the use of accessory respiratory muscles | From randomisation to discharge from intensive care or to Day 28
  Using the Patrick score (Score from 0 to 5)
Progression of dyspnoea | From randomisation to discharge from intensive care or to Day 28
  Assessed by the modified Borg scale (scale from 0 to 10)
Intensive care unit and/or continuous monitoring unit length of stay | From randomization until the date of discharge, assessed up to 28 days maximum
Intensive care unit and/or continuous monitoring unit length of stay or time to ICU discharge readiness | From randomization until the date of discharge OR ability to be discharged from intensive care, assessed up to 28 days maximum
  The ability to go out will be defined by the validation of all the items on the modified ability grid (score modified from Hiller et al. ; 28 items)

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Anh NAY, MD, Principal Investigator — CHRU Orléans
Locations (11):
- France (11):
  - Intensive care, University Hospital, Blois, Blois
  - Intensive care unit, University Hospital, Bourg-en-Bresse, Bourg-en-Bresse
  - Intensive care, University Hospital, Bourges, Bourges
  - Intensive care unit, University Hospital, Caen, Caen
  - Intensive care, University Hospital, Chartres, Chartres
  - Intensive care, University Hospital, Cholet, Cholet
  - Intensive care, University Hospital, Dax, Dax
  - Intensive care, University Hospital, Le Mans,, Le Mans
  - Intensive care, University Hospital, Orléans, Orléans
  - Intensive care, University Hospital, Tours, Tours
  - Intensive care unit, University Hospital, Vannes, Vannes